CLINICAL TRIAL: NCT01108471
Title: Study Comparing Non-Invasive Measurement of Hemoglobin (Using Pulse Co-Oximetry) With Laboratory Measurement in Patients Undergoing Elective Cesarean Delivery
Brief Title: Non-Invasive Measurement of Hemoglobin (Using Pulse Co-Oximetry) in Patients Undergoing Elective Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: SU-04082010-5622
Record Dates: First submitted 2010-04-14; First posted 2010-04-22 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Postpartum Hemorrhage
Keywords: cesarean section; hemoglobin; postpartum hemorrhage;
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We aim to assess a new pulse oximeter which measures continuous hemoglobin concentration (SpHb) in healthy patients undergoing elective Cesarean delivery (CS). This patient population often experiences significant blood loss during surgery, and measurements of surgical blood loss are often inaccurate. We will compare measurements of SpHb with estimated blood loss during the perioperative period, and laboratory measurements of hemoglobin at set time intervals during the perioperative and postoperative periods (to evaluate the accuracy of this device's ability to measure continuous SpHb).

DETAILED DESCRIPTION:
We hope that this pulse oximeter will provide important new information (SpHb) about hemoglobin measurement in patients undergoing elective CS, who may often experience significant blood loss and postpartum anemia in the perioperative period. The measurement of perioperative blood loss is often inaccurate, and formal measurements of hemoglobin levels are often associated with time delays, especially in the setting of ongoing acute blood loss. We hope that this device will provide accurate continuous data of hemoglobin in this patient population, which may prove to be a significant advance in patient monitoring in this patient population. Probes for SpHb measurement will be provided by Masimo Corporation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy term (> 37 weeks gestation)
2. ASA 1 and 2 pregnant patients undergoing elective uncomplicated Cesarean delivery under neuraxial anesthesia
3. Age 18-40 yrs

Exclusion Criteria:

1. Patients with abnormal Hemoglobin disorders.
2. Patients with hyperbilirubinemia.
3. Patients who are smokers.
4. Patients with peripheral vascular disease or conditions affecting vascularity of the digits.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy pregnant patients undergoing elective cesarean delivery under neuraxial anesthesia
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Total perioperative blood loss | Measured at the end of surgery (time frame cannto be specificied prior to study but estimated to be 60-90 mins)
  The total estimated blood loss will be assessed at the end of the surgical period. This period is estimated to be 60-90 mins. We will record the time duration of surgery for all patients in the study.
maternal SpHb | SpHb measurements will be measured at the following timepoints:prior to surgery,continuously during the intraoperative period; within 10 minutes of completion of surgery; at 4hr, 24hr, and 48 hr following completion of surgery
maternal venous hemoglobin measurements | Maternal venous hemoglobin measurements will be performed at the following timepoints: prior to surgery, within 10 minutes of completion of surgery, 24 hr following completion of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alex James Butwick, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Butwick A, Hilton G, Carvalho B. Non-invasive haemoglobin measurement in patients undergoing elective Caesarean section. Br J Anaesth. 2012 Feb;108(2):271-7. doi: 10.1093/bja/aer373. Epub 2011 Nov 23. PMID 22116296